CLINICAL TRIAL: NCT01960998
Title: Perioperative Post-Prostatectomy Incontinence Home Telehealth Program
Acronym: ProsTel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Emory University (Other); University of Pennsylvania (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1059-R
Record Dates: First submitted 2013-10-04; First posted 2013-10-11 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence; Prostate Cancer
Keywords: radical prostatectomy; urinary incontinence; prostate cancer; telehealth; pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Perioperative Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth with Pelvic Floor Muscle Training (Experimental): Participants in this group will participate in an evidence-based pelvic floor muscle training program that has been adapted to telehealth format. Training is begun 1 month before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively. In addition to the pelvic floor muscle training, content will also include general perioperative care; wetness, odor and skin care management; and outcome measures.
  Interventions: Behavioral: Pelvic Floor Muscle Training; Behavioral: Perioperative Care and Wetness Management
- Telehealth without Pelvic Floor Muscle Training (Active Comparator): Participants in this group will receive a telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 3 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
  Interventions: Behavioral: Perioperative Care and Wetness Management

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — Evidence-based pelvic floor muscle training program that has been adapted to telehealth format. Training is begun 2-4 weeks before surgery and continued 2 months after surgery. Content is accessed in daily 10-minute sessions on a secure website
  Arms: Telehealth with Pelvic Floor Muscle Training
Behavioral: Perioperative Care and Wetness Management — Telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.

SUMMARY:
Many men develop urine leakage after prostate cancer surgery. Usually it is temporary, but pelvic floor muscle training and exercise (including urine control strategies) have been shown to reduce the time to regaining urine control. This study tests an evidence-based, pelvic floor muscle training program that has been adapted to telehealth format and pilot tested in a VA-funded pilot/developmental trial. Training is begun 1-4 weeks before surgery and continued 6 months after surgery. Content is accessed on a secure website in daily 10-minute sessions which transition to weekly sessions for post-operative months 3-6. In the investigators' pilot study, Veterans reported that they appreciated receiving the training in the privacy of their homes, enjoyed the interactive style of the learning experience, and felt better prepared to deal with urine leakage and empowered with new knowledge and skills to help themselves. Content for both control and treatment groups includes general information about prostate cancer; perioperative care; wetness, odor and skin care management. The treatment group will ALSO receive pelvic floor muscle training and bladder control strategies. Outcomes are measured with brief validated questions administered by the telehealth platform, and again at 9 and 12 months by mailed questionnaire or the telehealth platform.

DETAILED DESCRIPTION:
Many men develop urine leakage after radical prostatectomy. Usually it is temporary, but pelvic floor muscle training including bladder control strategies has been shown to reduce the severity of incontinence and reduce the time to regaining continence. This study will test an evidence-based pelvic floor muscle training program that has been adapted to telehealth format and pilot tested in a VA-funded pilot/developmental trial. Training is begun 1-4 weeks before surgery and continued 6 months after surgery. Content is accessed on a secure website in daily 10-minute sessions which transition to weekly sessions for post-operative months 3-6. In the investigators' pilot study, Veterans reported that they appreciated receiving the training in the privacy of their homes, enjoyed the interactive style of the learning experience, and felt better prepared to deal with urine leakage and empowered with new knowledge and skills to help themselves.

This study is a randomized, controlled trial of the telehealth-delivered, evidence-based, intervention developed in the pilot/developmental study. Participants will be randomized 1:1 to treatment or to a control group. Content for both control and treatment groups includes general information about prostate cancer; perioperative care; wetness, odor and skin care management. The treatment group will ALSO receive pelvic floor muscle training and bladder control strategies. Outcomes are measured with brief validated questions administered by the telehealth platform, and again at 9 and 12 months by mailed questionnaire or the telehealth platform.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a radical prostatectomy for treatment of prostate cancer and enrolled at the Birmingham, Philadelphia, or Atlanta VA Medical Centers or the affiliated University Medical Centers
* Ability to read English.
* Internet access

Exclusion Criteria:

* Urinary Incontinence in the 6 months prior to prostate cancer surgery (other than post-void dribbling)
* Less than 1 week before surgery

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men planning surgery for prostate cancer
Enrollment: 245 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Burgio, PhD MA BA, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 245 participants were enrolled in the trial, but only 197 received the assigned intervention. 9 did not have the planned prostatectomy; 39 never started the assigned intervention.
Period: Overall Study
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Started | 101 | 96
Completed | 90 | 85
Not Completed | 11 | 11
Not completed — Lost to Follow-up | 3 | 7
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — lost computer access | 0 | 1

BASELINE CHARACTERISTICS:
Population: 245 participants were enrolled in the trial, but only 197 received the assigned intervention. 9 did not have the planned prostatectomy; 39 never started the assigned intervention.
Groups:
- Telehealth With Pelvic Floor Muscle Training: Participants in this group will participate in an evidence-based pelvic floor muscle training program that has been adapted to telehealth format. Training is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively. In addition to the pelvic floor muscle training, content will also include general perioperative care; wetness, odor and skin care management; and outcome measures.
  Pelvic Floor Muscle Training: Evidence-based pelvic floor muscle training program that has been adapted to telehealth format. Training is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in daily 10-minute sessions on a secure website
  Perioperative Care and Wetness Management: Telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
- Telehealth Without Pelvic Floor Muscle Training: Participants in this group will receive a telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
  Perioperative Care and Wetness Management: Telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
- Total: Total of all reporting groups
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (7.8) | 61.7 (7.1) | 61.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 122 | 123 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 122 | 121 | 243
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 27 | 65
  White | 82 | 95 | 177
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 122 | 123 | 245
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is a weight-to-height ratio used as an indicator of obesity and underweight. It is calculated by dividing an individual's weight in kilograms by the square of their height in meters.
  kg/m^2 | 28.2 (4.61) | 29.6 (4.54) | 28.9 (4.6)
Education [Count of Participants; unit: Participants]
  < High school | 1 | 2 | 3
  HS or GED | 39 | 36 | 75
  College or beyond | 82 | 85 | 167
Employment [Count of Participants; unit: Participants]
  Employed | 69 | 75 | 144
  Retired, disabled, or unemployed | 53 | 48 | 101
Living situation [Count of Participants; unit: Participants]
  Live alone | 14 | 10 | 24
  Live with family | 104 | 109 | 213
  Other | 4 | 4 | 8
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 14 | 9 | 23
  Former smoker | 46 | 42 | 88
  Never smoked | 62 | 72 | 134
Degenerative disc disease [Count of Participants; unit: Participants]
  Don't know | 1 | 0 | 1
  No | 103 | 96 | 199
  Yes | 18 | 27 | 45
Asthma, COPD [Count of Participants; unit: Participants]
  No | 108 | 113 | 221
  Yes | 14 | 10 | 24
Heart failure [Count of Participants; unit: Participants]
  No | 121 | 120 | 241
  Yes | 1 | 3 | 4
Diabetes [Count of Participants; unit: Participants]
  No | 98 | 109 | 207
  Yes | 24 | 14 | 38
Neurological disease [Count of Participants; unit: Participants]
  No | 119 | 120 | 239
  Yes | 3 | 3 | 6
Stroke or TIA [Count of Participants; unit: Participants]
  No | 117 | 121 | 238
  Yes | 5 | 2 | 7
Depression [Count of Participants; unit: Participants]
  No | 103 | 102 | 205
  Yes | 19 | 21 | 40
Anxiety [Count of Participants; unit: Participants]
  No | 111 | 102 | 213
  Yes | 10 | 21 | 31
  Missing | 1 | 0 | 1
Prostate specific antigen (PSA), ng/mL [Count of Participants; unit: Participants]
  < 10 | 3 | 8 | 11
  > or +10 | 119 | 115 | 234
Gleason score [Count of Participants; unit: Participants] — The Gleason score is used to describe prostate cancer cells based on pathologist examination of a biopsy sample. The cells are graded on a scale of 1 to 5, with Grade 1 cells resembling normal prostate tissue. Gleason scores usually range from 6 to 10. A Gleason score of 6 is low grade, 7 is intermediate grade, and 8 to 10 is high grade cancer.
  Participants
    < 7 | 32 | 36 | 68
    > or =7 | 90 | 87 | 177
Surgical approach [Count of Participants; unit: Participants]
  Retropubic | 102 | 97 | 199
  Perineal | 8 | 16 | 24
  Missing | 12 | 10 | 22
Surgical technique [Count of Participants; unit: Participants]
  Open | 5 | 4 | 9
  Robotic | 106 | 111 | 217
  Missing | 11 | 8 | 19
Neurovascular bundle sparing [Count of Participants; unit: Participants] — The neurovascular bundles lie postero-laterally to the prostate and are typically spared during prostatectomy to preserve sexual function. A "nerve-sparing" procedure involves dissecting the nerve bundle off the side of the prostate.
  Participants
    Both spared | 93 | 99 | 192
    One spared | 8 | 4 | 12
    None spared | 7 | 4 | 11
    Missing | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time to Continence
Description: Time to continence was based on the time point at which participants reported no urinary incontinence on the International Consultation on Incontinence (ICI) Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF). ICIQ-UI SF is one of a series of ICI questionnaires that have been meticulously developed and tested. The ICIQ-UI SF is a brief (4 items), reliable (Cronbach's alpha = 0.95), questionnaire that quantifies both symptom burden and impact of incontinence and has been validated in men and women. It was administered weekly during the 6 months after surgery. Scores range from 0-21; higher scores indicate worse condition.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Telehealth With Pelvic Floor Muscle Training: Participants in this group participated in an evidence-based pelvic floor muscle training program that was adapted to telehealth format. Training was begun 1-4 weeks before surgery and continued 2 months after surgery. Content was accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively. In addition to the pelvic floor muscle training, content also included general perioperative care; wetness, odor and skin care management; and outcome measures.
- Telehealth Without Pelvic Floor Muscle Training: Participants in this group received a telehealth program that included general perioperative care; wetness, odor and skin care management; and outcome measures. The program was begun 1-4 weeks before surgery and continued 2 months after surgery. Content was accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 96
weeks | NA [NA to NA] — Median survival time exceeded the observation period of 12 months in the telehealth group | NA [NA to NA] — Median survival time exceeded the observation period of 12 months in the no telehealth group
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.22, Log Rank — P value not adjusted for multiple comparisons; Data were not collected beyond the 12-month follow up, at which point fewer than 50% of participants in both groups had achieved continence. Thus, their time to continence could not be determined and the medians could not be calculated

2. Secondary Outcome: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) Total Score
Description: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form total score. Scores range from 0-21; higher scores indicate worse condition.
Time Frame: 6 months, 9 months, 12 months
Population: Two individuals were missing all outcome measures; data for these two participants were not imputed and were not included in the analysis, resulting in 94 individuals analyzed in the Telehealth without Pelvic Floor Muscle Training group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Telehealth With Pelvic Floor Muscle Training: Participants in this group will participate in an evidence-based pelvic floor muscle training program that has been adapted to telehealth format. Training is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively. In addition to the pelvic floor muscle training, content will also include general perioperative care; wetness, odor and skin care management; and outcome measures.
- Telehealth Without Pelvic Floor Muscle Training: Participants in this group will receive a telehealth program that includes include general perioperative care; wetness, odor and skin care management; and outcome measures. The program is begun 1-4 weeks before surgery and continued 2 months after surgery. Content is accessed in 10-minute sessions on a secure website - daily preoperatively and for the first 2 months post-operatively, then weekly until 6 months post-operatively.
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
score on a scale
  6 months | 7.1 (4.3) | 7.0 (4.4)
  9 months | 6.2 (3.9) | 6.7 (5.1)
  12 months | 5.9 (4.1) | 6.0 (4.7)
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.70, ANCOVA — P values were not corrected for multiple testing; Baseline score was included as a covariate in analysis; Mean values for the telehealth and no telehealth groups on the ICIQ-SF are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean ICIQ-SF score in the no telehealth group at 6 months was 7.0 (standard deviation 4.4) and in the telehealth group was 7.1 (SD 4.3). Analysis of covariance (ANCOVA) was performed with each of the 10 imputations, adjusting for baseline ICIQ-SF score, and p values were combined using the Rubin-Licht method

3. Secondary Outcome: Expanded Prostate Cancer Index Urinary Incontinence Subscale (EPIC-UI)
Description: This measure, validated as a stand-alone assessment, consists of 4 questions from the full Expanded Prostate Cancer Index (EPIC), a health-related quality of life assessment tool. The EPIC was developed based on advice from an expert panel and prostate cancer survivors, expanding the 20-item University of California - Los Angeles Prostate Cancer Index. Scores range from 0-100; higher scores indicate worse condition.
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
score on a scale
  6 months | 63.9 (22.1) | 63.5 (24.1)
  9 months | 67.7 (21.2) | 65.1 (26.2)
  12 months | 70.4 (20.4) | 68.0 (25.3)
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.70, ANCOVA — P values were not adjusted for multiple comparisons; Mean values for the telehealth and no telehealth groups on the EPIC-UI are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean EPIC-UI score in the no telehealth group at 6 months was 63.5 (standard deviation 24.1) and in the telehealth group was 63.9 (SD 22.1). Analysis of covariance (ANCOVA) was performed with each of the 10 imputations, adjusting for baseline EPIC-UI score, and p values were combined using the Rubin-Licht method

4. Secondary Outcome: Incontinence Impact Questionnaire - Short Form (IIQ-SF)
Description: This measure, validated in men with post-prostatectomy incontinence, measures the impact of incontinence on regular activities. It is a condition-specific quality of life measure that has been widely used in incontinence clinical trials. There are seven items. Response options are: "not at all," "slightly," "moderately," "greatly." Scores range from 0-100; higher scores indicate greater impact.
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
score on a scale
  6 months | 19.4 (22.4) | 22.3 (24.1)
  9 months | 15.2 (21.4) | 19.3 (24.9)
  12 months | 13.5 (20.7) | 16.5 (23.7)
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.46, t-test, 2 sided — P values not adjusted for multiple comparisons; Mean values for the telehealth and no telehealth groups on the IIQ are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean IIQ score in the no telehealth group at 6 months was 22.3 (standard deviation 24.1) and in the telehealth group was 19.4 (SD 22.4). Two-sample t-tests were performed with each of the 10 imputations, and p values were combined using the Rubin-Licht method

5. Secondary Outcome: International Prostate Symptom Scale - Quality of Life Question
Description: Validated single question: "If you were to spend the rest of your life with your urinary problem the way it is now, how would you feel about that?" Response options: delighted, pleased, mostly satisfied, mixed (about equally satisfied and dissatisfied), mostly dissatisfied, unhappy, terrible.
Time Frame: 6 months, 9 months, 12 months
Population: In both arms, the Outcome Measure Data Table reflects the average frequencies across 10 multiple imputations, so the sum of individual frequencies may not exactly equal the total number of participants due to rounding. Two individuals were missing all outcome measures; their data were not imputed and were not included in the analysis, resulting in 94 individuals analyzed in the Telehealth without Pelvic Floor Muscle Training group.
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months Delighted/Pleased | 21 | 30
  6 months Mostly satisfied | 27 | 21
  6 months Mixed | 27 | 18
  6 months Mostly dissatisfied | 13 | 11
  6 months Unhappy/Terrible | 14 | 14
  9 months Delighted/Pleased | 36 | 32
  9 months Mostly satisfied | 22 | 27
  9 months Mixed | 20 | 9
  9 months Mostly dissatisfied | 12 | 10
  9 months Unhappy/Terrible | 11 | 16
  12 months Delighted/Pleased | 41 | 39
  12 months Mostly satisfied | 28 | 25
  12 months Mixed | 17 | 12
  12 months Mostly dissatistied | 9 | 8
  12 months Unhappy/Terrible | 6 | 10
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.63, Chi-squared, Corrected — P values were not corrected for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the Quality of Life question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 31.4% (Delighted/Pleased), 22.8% (Mostly Satisfied), 19.4% (Mixed), 12.0% (Mostly Dissatisfied), and 14.4% (Unhappy/Terrible) and in the telehealth group were 20.8%, 26.3%, 26.3%, 12.6%, and 14.0%, respectively. Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 5 levels of the IPSS Quality of Life question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

6. Secondary Outcome: Patient Satisfaction Question (PSQ)
Description: Patient's rating of satisfaction (Completely satisfied, Somewhat satisfied, Not at all satisfied)
Time Frame: 6 months, 9 months, 12 months
Population: Two individuals were missing all outcome measures; data for these two participants were not imputed and were not included in the analysis, resulting in 94 individuals analyzed in the Telehealth without Pelvic Floor Muscle Training group. The frequencies for both Telehealth With and Without Pelvic Floor Muscle Training were calculated across 10 multiple imputations and rounded to the nearest whole number, so sum of individual categories (102) does not equal overall number of participants (101).
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: Completely satisfied | 35 | 48
  6 months: Somewhat satisfied | 61 | 38
  6 months: Not at all satisfied | 5 | 8
  9 months: Completely satisfied | 44 | 46
  9 months: Somewhat satisfied | 53 | 37
  9 months: Not at all satisfied | 4 | 11
  12 months: Completely satisfied | 54 | 50
  12 months: Somewhat satisfied | 42 | 34
  12 months: Not at all satisfied | 5 | 10
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.04, Chi-squared, Corrected — P values were not corrected for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the Patient Satisfaction question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 51.0% (Completely Satisfied), 40.2% (Somewhat Satisfied), and 8.7% (Not at All Satisfied) and in the telehealth group were 34.8%, 59.9%, and 5.3%, respectively (frequencies to not add to exactly 100% due to rounding). Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 3 levels of the Patient Satisfaction question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

7. Secondary Outcome: Estimated Percent Improvement (EPI)
Description: Participant self-report of perceived percent improvement from 0% to 100%
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
percent improvement
  6 months | 69.6 (29.6) | 65.1 (34.5)
  9 months | 76.0 (26.2) | 72.6 (31.8)
  12 months | 77.4 (28.7) | 75.7 (28.8)
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.67, t-test, 2 sided — P values not adjusted for multiple comparisons; Mean values for the telehealth and no telehealth groups on the Estimated Percent Improvement (EPI) are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean EPI score in the no telehealth group at 6 months was 65.1 (standard deviation 34.5) and in the telehealth group was 69.6 (SD 29.6). Two-sample t-tests were performed with each of the 10 imputations, and p values were combined using the Rubin-Licht method

8. Secondary Outcome: Global Perception of Improvement (GPI)
Description: Participant's global perception of their improvement (Much better, Better, About the same, Worse, Much worse)
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: Much better | 39 | 43
  6 months: Better | 41 | 29
  6 months: About the same | 15 | 16
  6 months: Worse | 3 | 2
  6 months: Much worse | 3 | 4
  9 months: Much better | 41 | 43
  9 months: Better | 45 | 29
  9 months: About the same | 9 | 15
  9 months: Worse | 3 | 4
  9 months: Much worse | 3 | 3
  12 months: Much better | 51 | 43
  12 months: Better | 31 | 25
  12 months: About the same | 12 | 19
  12 months: Worse | 2 | 3
  12 months: Much worse | 5 | 4
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.65, Chi-squared, Corrected; Frequencies for the telehealth and no telehealth groups on the Global Perception of Improvement (GPI) question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 46.3% (Much Better), 30.7% (Better), 16.7% (About the Same), 2.3% (Worse), and 3.9% (Much Worse) and in the telehealth group were 38.3%, 41.1%, 15.3%, 2.9%, and 2.5%, respectively (frequencies to not add to exactly 100% due to rounding). Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 5 levels of the Global Perception of Improvement question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

9. Secondary Outcome: How Disturbing is Urine Leakage
Description: Single quality of life question: "How disturbing is the urine leakage problem to you?" (not at all, somewhat, or extremely disturbing)
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: Not at all | 39 | 41
  6 months: Somewhat | 54 | 42
  6 months: Extremely | 8 | 11
  9 months: Not at all | 42 | 42
  9 months: Somewhat | 53 | 45
  9 months: Extremely | 6 | 7
  12 months: Not at all | 43 | 49
  12 months: Somewhat | 51 | 34
  12 months: Extremely | 7 | 11
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.37, Chi-squared, Corrected — P values were not corrected for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the "How Disturbing is the Urine Leakage?" question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 43.5% (Not at All), 44.4% (Somewhat), and 12.1% (Extremely) and in the telehealth group were 38.9%, 53.2%, and 7.9% respectively. Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 3 levels of the "How Disturbing is the Urine Leakage?" question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

10. Secondary Outcome: Activity Restriction
Description: Single quality of life question: "How much does leakage of urine restrict your activities?" (not at all, some of the time, most of the time, all of the time).
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: Not at all | 57 | 48
  6 months: Some of the time | 34 | 34
  6 months: Most of the time | 4 | 7
  6 months: All of the time | 6 | 5
  9 months: Not at all | 70 | 63
  9 months: Some of the time | 25 | 23
  9 months: Most of the time | 1 | 4
  9 months: All of the time | 5 | 4
  12 months: Not at all | 74 | 65
  12 months: Some of the time | 19 | 17
  12 months: Most of the time | 4 | 7
  12 months: All of the time | 4 | 5
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.63, Chi-squared, Corrected — P values were not adjusted for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the Activity Restriction question relative to the expected frequencies question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 51.0% (Not at all), 36.5% (Some of the time), 7.2% (Most of the time), and 5.3% (All of the time) and in the telehealth group were 56.5%, 33.5%, 4.2%, and 5.8% respectively (frequencies to not add to exactly 100% due to rounding). Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 4 levels of the Activity Restriction question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

11. Secondary Outcome: Return to Work
Description: Single quality of life question: "Have you been able to return to work since your surgery?" (yes, no, retired or disabled)
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: Yes | 63 | 49
  6 months: No, not yet recovered from surgery | 3 | 5
  6 months: No, other reason | 1 | 2
  6 months: Retired or disabled | 34 | 38
  9 months: Yes | 62 | 55
  9 months: No, not yet recovered from surgery | 3 | 2
  9 months: No, other reason | 1 | 3
  9 months: Retired or disabled | 35 | 34
  12 months: Yes | 66 | 52
  12 months: No, not yet recovered from surgery | 3 | 4
  12 months: No, other reason | 1 | 2
  12 months: Retired or disabled | 31 | 36
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.71, Chi-squared, Corrected — P values not adjusted for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the Return to Work question relative to the expected frequencies question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 52.3% (Yes), 5.0% (No, not yet recovered from surgery), 1.9% (No, other reason), and 40.7% (Retired or disabled) and in the telehealth group were 62.3%, 3.5%, 0.8%, and 33.5% respectively (frequencies to not add to exactly 100% due to rounding). Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 4 levels of the Return to Work question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

12. Secondary Outcome: Resumption of Normal Activity
Description: Single quality of life question: "Have you been able to resume your usual activities since your surgery?" (yes, no)
Time Frame: 6 months, 9 months, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
Number analyzed (Participants) | 101 | 94
Participants
  6 months: None | 5 | 7
  6 months: Some | 23 | 28
  6 months: All | 73 | 59
  9 months: None | 4 | 5
  9 months: Some | 19 | 19
  9 months: All | 78 | 70
  12 months: None | 4 | 3
  12 months: Some | 16 | 17
  12 months: All | 81 | 74
Statistical Analysis 1: Comparison: Telehealth With Pelvic Floor Muscle Training vs Telehealth Without Pelvic Floor Muscle Training; Test type: Superiority; p = 0.41, Chi-squared, Corrected — P values not corrected for multiple comparisons; Frequencies for the telehealth and no telehealth groups on the Resumption of Normal Activities question relative to the expected frequencies question are presented above. Multiple imputation was performed to account for missing data, using the Multiple Imputation via Chained Equations (MICE) package in R. Across 10 imputations, the mean frequencies for the no telehealth group at 6 months were 7.4% (None), 29.8% (Some), 62.8% (All) and in the telehealth group were 4.9%, 23.0%, and 72.2% respectively (frequencies to not add to exactly 100% due to rounding). Chi-squared analysis with continuity correction was used to determine if there were differences in the observed frequencies between groups (telehealth versus no telehealth) across the 3 levels of the Resumption of Normal Activities question relative to the expected frequencies with each of the imputations, and p values were combined using the Enders (2001) method

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Telehealth With Pelvic Floor Muscle Training | Telehealth Without Pelvic Floor Muscle Training
All-Cause Mortality (participants affected / at risk) | 0/101 | 1/96
Serious Adverse Events (participants affected / at risk) | 0/101 | 1/96
Other Adverse Events (participants affected / at risk) | 0/101 | 1/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telehealth With Pelvic Floor Muscle Training (N=101) | Telehealth Without Pelvic Floor Muscle Training (N=96)
Death (General disorders) | 0 | 1 — Participant's wife informed the study coordinator that the participant had passed away, after the study coordinator attempted to contact the participant. The event was determined to be anticipated in an older adult and unrelated to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telehealth With Pelvic Floor Muscle Training (N=101) | Telehealth Without Pelvic Floor Muscle Training (N=96)
Complications of surgery (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT01960998/Prot_SAP_000.pdf